CLINICAL TRIAL: NCT03815890
Title: Pre-operative Phase II Trial for Breast Cancer With Nivolumab in Combination With Novel IO (BELLINI Trial)
Brief Title: Pre-operative Trial for Breast Cancer With Nivolumab in Combination With Novel IO
Acronym: BELLINI
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M18BEL
Record Dates: First submitted 2018-12-13; First posted 2019-01-24 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Breast Cancer
Keywords: pre-operative; triple negative and Luminal B; resectable, stage I-III
MeSH Terms: conditions — Breast Neoplasms | interventions — Nivolumab; Ipilimumab

STUDY DESIGN:
Intervention Model Description: Separate cohorts will be opened in this trial. LumB and TNBC tumors will be divided in separate cohorts.More cohorts, e.g. combining nivolumab and novel IO, can open after the start of this trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1A; LumB (Experimental): Nivolumab
  Interventions: Drug: Nivolumab
- 1B; TNBC (Experimental): Nivolumab
  Interventions: Drug: Nivolumab
- 2A; LUMB (Experimental): Nivolumab and ipilimumab
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- 2B; TNBC (Experimental): Nivolumab and ipilimumab
  Interventions: Drug: Nivolumab; Drug: Ipilimumab
- 3B; TNBC, High TIL (Experimental): Nivolumab and ipilimumab
  Interventions: Drug: Nivolumab; Drug: Ipilimumab

INTERVENTIONS:
Drug: Nivolumab — 2 courses 240 mg flat dose
Drug: Ipilimumab — single dose ipilimumab (1mg/kg) at day 1
  Arms: 2A; LUMB; 2B; TNBC
Drug: Ipilimumab — two courses ipilimumab (1mg/kg) at day 1 and 21
  Arms: 3B; TNBC, High TIL

SUMMARY:
To determine whether short-term pre-operative nivolumab either as monotherapy or in combination with low dose doxorubicin or novel IO combinations can induce immune activation in early BC.

DETAILED DESCRIPTION:
The investigators aim to test the activity of nivolumab monotherapy in primary breast tumors in a pre-operative window of opportunity trial. As the data of the investigators generated in the TONIC trial (metastatic TNBC) indicate that low dose doxorubicin may 'prime' the tumor microenvironment (TME) resulting in higher response rates on nivolumab, in addition, cohorts for treatment with nivolumab plus low dose doxorubicin will be opened. Given the emerging data on other immunomodulatory strategies, this platform study allows opening additional cohorts for promising novel immune-oncology (IO) drugs for which a strong efficacy signal has been seen without drug safety issues. The investigators will study the TME and systemic host factors with specific emphasis on immunosuppressive processes that can potentially be targeted by novel IO agents to further optimize BC immunotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* 18 years or older at moment of inclusion;
* Female gender;
* WHO performance status 0 or 1;
* Resectable primary breast cancer stage I-III. Nodal status must be examined by ultrasound, fine needle aspiration, sentinel node biopsy, or FDG-PET scan.
* The tumors must be:

  * at least 10 mm (minimum cT1c) as determined by MRI
  * TNBC defined as ER<10%, HER2-negative OR luminal B defined as ER≥10%, HER2-negative with either Ki67≥20% or PR =<20% OR grade 3. HER2 negative is defined as an IHC score of <2 or 2+ with a negative ISH.
  * For TNBC patients: TIL≥5%
  * For LumB breast cancer patients: TIL≥1%
  * For cohort 3B: N0 status, TN and TIL ≥50%
  * For cohort 4B: N0 status, TNBC and TIL 30-49%
  * For cohort 5B: N0 status, TNBC and TIL ≥50% ● Patients with multifocal/multicentric breast cancer are eligible if triple negative breast cancer histology as well as sufficient TIL percentages (30-49% in cohort 4B, ≥50% in cohort 5B) have been confirmed in all tumor lesions.

Exclusion Criteria:

* evidence or suspicion of metastatic disease. Evaluation of the presence of distant metastases may include chest X-ray, liver ultrasound, isotope bone-scan, CT-scan of chest and abdomen and/or FDG-PET scan, according to local procedures;
* evidence of a concurrent contralateral or ipsilateral second primary infiltrating breast cancer. Evaluation of the presence of a concurrent second primary breast cancer may include mammography, breast ultrasound and/or MRI breast;
* other malignancy except carcinoma in situ and basal-cell and squamous carcinoma of the skin, unless the other malignancy was treated ≥5 years ago with curative intent without the use of chemotherapy or radiotherapy
* previous radiation therapy or chemotherapy;
* prior treatment with checkpoint inhibitors (including anti- PD1, -PD-L1, -CTLA-4);
* concurrent anti-cancer treatment, neoadjuvant therapy or another investigational drug;

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-10-04 (Actual); Primary Completion 2031-01-01 (Estimated); Study Completion 2033-01-01 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response rate per cohort, | up to 3 weeks after surgery, an average of 6 months
  number of patients with no residual invasively growing tumor cells detected by microscopic examination in breast and axilla

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events according to NCI Common Toxicity Criteria version 5.0 | up to 3 weeks after surgery, an average of 6 months
  Adverse events in all regimens will be graded according to NCI Common Toxicity Criteria version 5.0.
Radiological response rate | At 4 weeks
  The percentage of patients having a complete response, partial response or stable disease per cohort assessed by MRI
Immune activation after pre-operative nivolumab, either as monotherapy or in combination with ipilimumab or relatlimab or novel IO combinations. | within 6 months after surgery
  Immune activation is defined as either a 2-fold increase in tumor-associated CD8 after pre-operative immunotherapy; and/or a 2-fold increase expression of genes induced by IFNy (determined using mRNA expression levels)

CONTACTS AND LOCATIONS:
Overall Officials: M Kok, MD, Principal Investigator — NKI-AvL
Locations (1):
- NKI-AVL, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
to be determined

REFERENCES:
- [Derived] Nederlof I, Isaeva OI, de Graaf M, Gielen RCAM, Bakker NAM, Rolfes AL, Garner H, Boeckx B, Traets JJH, Mandjes IAM, de Maaker M, van Brussel T, Chelushkin M, Champanhet E, Lopez-Yurda M, van de Vijver K, van den Berg JG, Hofland I, Klioueva N, Mann RM, Loo CE, van Duijnhoven FH, Skinner V, Luykx S, Kerver E, Kalashnikova E, van Dongen MGJ, Sonke GS, Linn SC, Blank CU, de Visser KE, Salgado R, Wessels LFA, Drukker CA, Schumacher TN, Horlings HM, Lambrechts D, Kok M. Neoadjuvant nivolumab or nivolumab plus ipilimumab in early-stage triple-negative breast cancer: a phase 2 adaptive trial. Nat Med. 2024 Nov;30(11):3223-3235. doi: 10.1038/s41591-024-03249-3. Epub 2024 Sep 16. PMID 39284953